CLINICAL TRIAL: NCT00864227
Title: A Multi-Center, Phase II Trial of Non-Myeloablative Conditioning (NST) and Transplantation of Umbilical Cord Blood (UCB) From Unrelated Donors in Patients With Hematologic Malignancies (BMT CTN #0604)
Brief Title: Evaluating the Safety and Effectiveness of an Umbilical Cord Blood Stem Cell Transplant (BMT CTN 0604)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0604; U01HL069294 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse
Keywords: Acute Lymphoblastic Leukemia/Lymphoma; Acute Myelogenous Leukemia; Mantel-Cell Lymphoma; Hematopoietic Transplant; Umbilical Cord Blood (UCB); Non-Myeloablative Transplant
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical Cord Blood Transplantation (Experimental): Participants will receive a double unit Hematopoietic Umbilical Cord Blood Stem Cell Transplantation using a non-myeloablative preparative regimen, GVHD prophylaxis.
  Interventions: Biological: Hematopoietic Umbilical Cord Blood Stem Cell Transplantation; Biological: GVHD prophylaxis

INTERVENTIONS:
Biological: Hematopoietic Umbilical Cord Blood Stem Cell Transplantation — The transplant preparative regimen is listed below. The - sign is the number of days before the transplant.
  * Fludarabine: 40 mg/m^2 intravenously (IV) on Days -6, -5, -4, -3, and -2
  * Cyclophosphamide: 50 mg/kg IV on Day -6
  * Total body irradiation: 200 centigray (cGy) on Day -1
Biological: GVHD prophylaxis — GVHD prophylaxis regimen will consist of:
  * Cyclosporine: beginning on Day -3 with the dose adjusted to maintain a level of 200-400 mg/mL
  * MMF: 1 gram IV three times a day (TID) if greater than 50 kg, or 15 mg/kg IV TID if less than 50 kg beginning on Day -3; continued until Day 30 or 7 days after engraftment, whichever day is later
  Day 0 is the day of the infusion of the umbilical cord blood graft units, which will be obtained from partially HLA-matched unrelated donors.
  Beginning on Day 1, participants will receive G-CSF 5 mcg/kg/day until absolute neutrophil count (ANC) is greater than or equal to 2,000/mm^3 for three consecutive measurements, each on different days.

SUMMARY:
A bone marrow transplant, which is a type of stem cell transplant, is a treatment option for people with leukemia or lymphoma. Recently, stem cell transplants using umbilical cord blood have become a treatment option for people with these types of cancers. This study will evaluate the effectiveness of a stem cell transplant using umbilical cord blood, along with lower doses of chemotherapy, to treat people with leukemia or lymphoma.

DETAILED DESCRIPTION:
Leukemia and lymphoma are types of blood cancers. Chemotherapy is a common treatment option for people with these types of cancers, but if the cancer does not respond well to chemotherapy, or if the cancer returns, people may need to consider other options. A bone marrow transplant, which is a type of stem cell transplant in which healthy bone marrow is donated to a patient by a related or unrelated donor, is commonly used to treat leukemia and lymphoma. Recently, stem cell transplants using umbilical cord blood have become a viable option to treat these types of cancers. Traditionally, umbilical cord blood, which is the blood left over in the placenta after a baby is born, has been disposed of with the placenta. However, over the past few years, doctors have begun to collect and freeze the umbilical cord blood cells so that they may be used in stem cell transplant procedures at a later time.

Typically, people who are undergoing a stem cell transplant receive high doses of chemotherapy before the transplant to prepare their bodies to accept the donor stem cells. In this study, participants will undergo a new type of stem cell transplant called a nonmyeloablative transplant, which is a reduced intensity method of transplantation that does not require high doses of chemotherapy. The purpose of the study is to examine the safety and effectiveness of a nonmyeloablative stem cell transplant that uses umbilical cord blood as a treatment option for people with leukemia or lymphoma.

This study will enroll people with leukemia or lymphoma. Participants will be admitted to the hospital and will first receive a type of chemotherapy called cyclophosphamide, which will be given intravenously on the sixth day before the transplant. In addition, another type of chemotherapy, fludarabine, will be given intravenously each day for 5 days before the transplant. Three days before the transplant, participants will receive cyclosporine and mycophenolate mofetil (MMF), to help prevent the body from rejecting the stem cells and to help decrease the risk of developing a complication called graft-versus-host-disease (GVHD), which is an attack by the donor cells on the body's normal tissues. Some participants may receive tacrolimus instead of cyclosporine. After 6 days, participants will receive a small dose of radiation. The next day, participants will undergo the umbilical cord blood stem cell transplant.

Participants will remain in the hospital for approximately 2 to 3 months total, but possibly longer if there are complications. Beginning on the first day after the transplant, participants will receive daily injections of a growth factor called granulocyte-colony stimulating factor (G-CSF), which is a natural protein that increases the white blood cell count; G-CSF will be continued until a participant's white blood cell count is normal again. Participants will continue to receive MMF for 30 days and cyclosporine or tacrolimus for 180 days after the transplant. While participants are in the hospital, blood samples will be collected regularly to evaluate the response and possible side effects to treatment, including GVHD. If necessary, participants will receive platelet and red blood cell transfusions. At follow-up study visits 6 months and 1 year after the transplant, blood samples will be obtained. Study researchers will keep track of participants' medical condition through phone calls or mailings to participants and their doctors once a year for the rest of the participants' lives.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 21 to 70 years old; participants 1 to 21 years old are also eligible if they are ineligible for BMT CTN #0501 (NCT00412360)
* Each unit must supply a minimum of 1.5 x 10^7/kg pre-cryopreserved nucleated cell dose
* Participants must have two partially human leucocyte antigen (HLA)-matched umbilical cord blood units. Each unit must match at a minimum of 4 of 6 at HLA-A, -B, -DRB1 loci with the recipient. This may include 0 to 2 antigen mismatches at each A or B (at the antigen level) or DRB1 (at the allele level) loci. Each unit must be a 4 to 6 HLA-A, B, and DRB1 antigen matched to each other, not necessarily at the same loci as with the recipient. All typing will be done using molecular typing. Though molecular level typing will be available, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1 for this study. An adult unrelated donor search is not required for a person to be eligible for this study if the clinical situation dictates an urgent transplant. Clinical urgency is defined as 6 to 8 weeks from referral to transplant center or low likelihood of finding a matched, unrelated donor.
* Must have received cytotoxic chemotherapy within 3 months of the consent date (measured from the start date of chemotherapy)
* Acute leukemias (includes T lymphoblastic lymphoma) in the second or subsequent complete remission (CR)
* Burkitt's lymphoma in the second or subsequent CR
* Lymphoma
* Patients with adequate physical function, as measured by the following:

  * Heart: left ventricular ejection fraction at rest greater than 35%, or shortening fraction greater than 25%
  * Liver: bilirubin less than or equal to 2.5 mg/dL and alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than or equal to five times the upper limit of normal
  * Kidney: serum creatinine within normal range for age, or if serum creatinine is outside the normal range for age, then kidney function (creatinine clearance or glomerular filtration rate (GFR) greater than 40 mL/min/1.73m^2
  * Lungs: forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and carbon monoxide diffusing capacity (DLCO) greater than 50% predicted (corrected for hemoglobin). If unable to perform pulmonary function tests, then oxygen (O2) saturation must be greater than 92% on room air.

Exclusion Criteria:

* Have an HLA-matched, related, or 7 or 8/8 HLA allele matched (HLA-A, -B, -Cw, -DRB1) related donor able to donate
* Had an autologous hematopoietic stem cell transplant in the 3 months before study entry
* Pregnant or breastfeeding
* Evidence of HIV infection or known HIV positive serology
* Current uncontrolled bacterial, viral, or fungal infection (i.e., currently taking medication with evidence of progression of clinical symptoms or radiologic findings)
* Prior allogeneic hematopoietic stem cell transplant
* History of primary idiopathic myelofibrosis

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research (CIBMTR), Medical College of Wisconsin
Locations (16):
- United States (16):
  - City of Hope National Medical Center, Duarte, California
  - University of Florida College of Medicine, Shands, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Dana-Farber Cancer Institute (DFCI), Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, Barnes Jewish Hospital, St Louis, Missouri
  - Weill Cornell Medical College, NY Presbyterian Hospital, New York, New York
  - Ohio State, Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University, Medical College of Virginia (MCV) Hospital, Richmond, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Findings will be published in a manuscript.

REFERENCES:
- [Result] Brunstein CG, Fuchs EJ, Carter SL, Karanes C, Costa LJ, Wu J, Devine SM, Wingard JR, Aljitawi OS, Cutler CS, Jagasia MH, Ballen KK, Eapen M, O'Donnell PV; Blood and Marrow Transplant Clinical Trials Network. Alternative donor transplantation after reduced intensity conditioning: results of parallel phase 2 trials using partially HLA-mismatched related bone marrow or unrelated double umbilical cord blood grafts. Blood. 2011 Jul 14;118(2):282-8. doi: 10.1182/blood-2011-03-344853. Epub 2011 Apr 28. PMID 21527516
- [Result] Eapen M, O'Donnell P, Brunstein CG, Wu J, Barowski K, Mendizabal A, Fuchs EJ. Mismatched related and unrelated donors for allogeneic hematopoietic cell transplantation for adults with hematologic malignancies. Biol Blood Marrow Transplant. 2014 Oct;20(10):1485-92. doi: 10.1016/j.bbmt.2014.05.015. Epub 2014 May 23. PMID 24862638

RESULTS

PARTICIPANT FLOW:
Groups:
- dUCB Transplant: Hematopoietic Umbilical Cord Blood Stem Cell Transplantation using a non-myeloablative preparative regimen.
Period: Overall Study
Arm/Group | dUCB Transplant
Started | 54
Completed | 50
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Disease Relapse/Progression | 3

BASELINE CHARACTERISTICS:
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Karnofsky Performance-status Score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    100% | 10
    90% | 30
    80% | 7
    70% | 2
    60% | 1
Primary Disease [Number; unit: participants]
  Acute Lymphoblastic Leukemia | 6
  Acute Myelogeneous Leukemia | 29
  Biphenotypic/Undifferentiated Leukemia | 1
  Burkitt's Lymphoma | 1
  Hodgkins Lymphoma | 5
  Large Cell Lymphoma | 3
  Marginal Zone B-cell Lymphoma | 1
  Follicular Non-Hodgkins Lymphoma | 4
HLA Typing Match Score - 1st Cord [Number; unit: participants] — Units must be HLA-matched at 4 of 6 HLA-A and B (intermediate resolution molecular typing) and DRB1 (high resolution molecular typing) with each other and 4 of 6 with the recipient.
  participants
    4/6 | 24
    5/6 | 21
    6/6 | 5
HLA Typing Match Score - 2nd Cord [Number; unit: participants] — Units must be HLA-matched at 4 of 6 HLA-A and B (intermediate resolution molecular typing) and DRB1 (high resolution molecular typing) with each other and 4 of 6 with the recipient.
  participants
    4/6 | 30
    5/6 | 17
    6/6 | 3
HLA Typing Match Score - 1st Cord to 2nd Cord [Number; unit: participants] — Units must be HLA-matched at 4 of 6 HLA-A and B (intermediate resolution molecular typing) and DRB1 (high resolution molecular typing) with each other and 4 of 6 with the recipient.
  participants
    4/6 | 35
    5/6 | 11
    6/6 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 180 Days From the Time of Transplant
Time Frame: Measured at Month 6 and Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
percentage of participants
  6 months | 73.5 [58.8 to 83.7]
  1 year | 54.0 [38.3 to 67.3]

2. Secondary Outcome: Neutrophil Recovery
Description: Neutrophil recovery is defined as achieving an absolute neutrophil count ≥ 500/mm3 for three consecutive measurements on different days.
Time Frame: Measured at Days 28, 56, 90, and 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
percentage of participants
  Day 28 | 86.0 [76.0 to 96.0]
  Day 56 | 94.0 [86.6 to 100.0]
  Day 90 | 94.0 [86.6 to 100.0]
  Day 100 | 94.0 [86.6 to 100.0]

3. Secondary Outcome: Primary Graft Failure
Description: Primary graft failure is defined as < 5% donor chimerism on all measurements prior to and day-100.
Time Frame: Measured at Day 100
Measure: Number; unit: participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
participants | 5

4. Secondary Outcome: Secondary Graft Failure
Description: Secondary graft failure is defined initial recovery followed by neutropenia with < 5% donor chimerism.
Time Frame: Measured at Day 100
Measure: Number; unit: participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
participants | 1

5. Secondary Outcome: Platelet Recovery to 20K
Description: Platelet recovery is defined as the first day of a minimum of three consecutive measurements on different days such that the patient has achieved a platelet count >20,000/mm3 with no platelet transfusions in the preceding seven days.
Time Frame: Measured at Days 56, 90, and 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
percentage of participants
  Day 56 | 70.0 [57.1 to 82.9]
  Day 90 | 82.0 [71.0 to 93.0]
  Day 100 | 82.0 [71.0 to 93.0]

6. Secondary Outcome: Donor Cell Engraftment
Description: Marrow or Blood Sample. Donor cell engraftment is defined as donor chimerism ≥ 5% on Day ≥ 56 after transplantation. Chimerism should be evaluated on Days ~28, ~56, ~180, and ~365 after transplantation. Chimerism may be evaluated in whole blood or mononuclear fraction.
Time Frame: Measured at Day 56
Measure: Number; unit: participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
participants
  Chimerism Performed | 36
  Donor Percentage >=95% | 30
  Donor Percentage 5%-95% | 6
  Donor Percentage <5% | 0

7. Secondary Outcome: Acute Graft-versus-host Disease (GVHD)
Time Frame: Measured at Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
percentage of participants
  Grade II-IV Acute GVHD | 40.0 [26.3 to 53.7]
  Grade III-IV Acute GVHD | 21.4 [5.9 to 36.9]

8. Secondary Outcome: Chronic GVHD
Time Frame: Measured at Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
percentage of participants | 25.3 [11.8 to 38.8]

9. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the minimum time interval to relapse/ recurrence/progression, to death or to last follow-up.
Time Frame: Measured at Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
percentage of participants | 45.7 [30.7 to 59.6]

10. Secondary Outcome: Treatment-related Mortality (TRM)
Time Frame: Measured at 6 months and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
percentage of participants
  6 months | 16.3 [5.9 to 26.7]
  1 year | 23.8 [11.3 to 36.3]

11. Secondary Outcome: Incidence of Infections
Description: Number of participants that experienced at least one infection.
Time Frame: Measured at Year 1
Measure: Number; unit: Infections
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
Infections
  1 Infection | 11
  2 Infections | 11
  3 Infections | 3
  4 Infections | 4
  5 Infections | 3
  6-10 Infections | 8
  >10 Infections | 1

12. Secondary Outcome: Platelet Recovery to 50K
Description: Platelet recovery is defined as the first day of a minimum of three consecutive measurements on different days such that the patient has achieved a platelet count >50,000/mm3 with no platelet transfusions in the preceding seven days.
Time Frame: Measured at Days 56, 90, and 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | dUCB Transplant
Number analyzed (Participants) | 50
percentage of participants
  Day 56 | 46.0 [31.9 to 60.1]
  Day 90 | 58.5 [44.4 to 72.6]
  Day 100 | 58.5 [44.4 to 72.6]

ADVERSE EVENTS:
Time Frame: 1-year post-transplant
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event.
Arm/Group | dUCB Transplant
Serious Adverse Events (participants affected / at risk) | 9/50
Other Adverse Events (participants affected / at risk) | 1/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dUCB Transplant (N=50)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Mechanical ventilation (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dUCB Transplant (N=50)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-01-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT00864227/Prot_SAP_ICF_001.pdf